CLINICAL TRIAL: NCT00201565
Title: Association Between Peripheral Artery Stiffness and Cardiovascular Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700336
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-03

CONDITIONS: Arteriosclerosis
Keywords: pulse wave velocity; cardiovascular disease
MeSH Terms: conditions — Arteriosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Arterial pulse wave velocity (PWV) is strongly correlated with atherosclerosis, and the PWV of carotid or femoral artery could predict the severity of arterial atherosclerosis. Because the measurement of PWV is noninvasive, it would serve as a good clinical and screen marker to evaluate the extent of atherosclerosis. The study uses self-made PWV measurement device to investigate the correlation of the PWV in the high cardiovascular risk population, and compare it with normal population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a high risk for cardiovascular disease

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Juey Jen Hwang, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Natinal Taiwan University Hospital, Taipei, Taiwan